CLINICAL TRIAL: NCT00478686
Title: A Retrospective Analysis of the Association of Dihydropyrimidine Dehydrogenase (DPYD) Variants With Toxicity Related to Capecitabine
Brief Title: Association of Dihydropyrimidine Dehydrogenase (DPYD) Variants With Toxicity Related to Capecitabine
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Myrexis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-1003
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Dihydropyrimidine Dehydrogenase; DPYD; DPYD Variants; Toxicity; Capecitabine; Xeloda
MeSH Terms: conditions — Breast Neoplasms | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 5 to 7.5 milliliter (mL) sample of blood. Alternatively, DNA will be extracted from 10um slices of formalin-fixed paraffin-embedded tissue from previously collected tumor tissue (from the time of the breast cancer diagnosis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Toxicity: Patients who experienced severe toxicity (at least one grade 4 side effect) with capecitabine chemotherapy
  Interventions: Procedure: Phlebotomy
- Dose-Limiting Toxicity: Patients who experienced dose-limiting toxicity (at least one grade 3, or recurrent grade 2, side effect)with capecitabine chemotherapy
  Interventions: Procedure: Phlebotomy
- Low/No Toxicity: Patients who have experienced low/no toxicity (none or only side effects at grade 1 & 2) with capecitabine chemotherapy.
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — 5 to 7.5 milliliter (mL) Blood Sample

SUMMARY:
The goal of this laboratory research study is to identify possible differences in a gene among patients with breast cancer that cannot be treated by surgery. Researchers want to find out if differences in this gene may increase the risk of side effects from capecitabine.

DETAILED DESCRIPTION:
If you agree to take part in this study, 1 blood sample (about 2 tablespoons) will be drawn for use in genetic research.

If you are unable to provide a blood sample, researchers will collect leftover tissue samples from your previously collected tumor tissue (from the time of the breast cancer diagnosis). The tumor samples will be used for genetic research.

After the blood draw or tissue collection, your participation in this study will be over.

The blood samples for the genetic research will be stored at Myriad Laboratories. Before your blood and/or tissue is sent to Myriad Laboratories for banking, your name and any personal identifying information will be coded to protect your privacy. M. D. Anderson will not have oversight of any leftover tissue and/or blood that will be banked by Myriad Laboratories for additional research.

This is an investigational study. Up to 210 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be registered for protocol ID 01-580 and only patients who were randomized to receive capecitabine will be included in the study.
2. Patients must sign an informed consent for this protocol.

Exclusion Criteria:

1) There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast cancer who experienced toxicity/side effects related to capecitabine chemotherapy.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2007-05-23 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Incidence of DPYD variants in patients | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org